CLINICAL TRIAL: NCT07133464
Title: CDH1-associated Blepharocheilodontic Syndrome Registry
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Maegan Roberts, Assistant Professor, Ohio State University
Other Study IDs: STUDY20250005
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Blepharocheilodontic Syndrome
Keywords: CDH1; Blepharocheilodontic Syndrome; Blepharocheilodontic; BCDS; CDH1-associated Blepharocheilodontic Syndrome; ectodermal dysplasia; cleft lip and palate; eyelid malformations
MeSH Terms: conditions — Blepharo-cheilo-dontic syndrome; Ectodermal Dysplasia; Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals identified as having a CDH1 variant and features of blepharocheilodontic syndrome

SUMMARY:
The aim of the CDH1-associated Blepharocheilodontic Syndrome (BCDS) registry is to better characterize the clinical features of this condition and exploring whether CDH1 variants linked to BCDS may also increase cancer risk.

DETAILED DESCRIPTION:
Blepharocheilodontic Syndrome (BCDS) is a rare genetic disorder characterized by cleft lip and/or palate (CL/P), eyelid malformations, and features suggestive of ectodermal dysplasia. Variants in the CDH1 gene, which encodes the cell adhesion protein E-cadherin, have been implicated in BCDS. Functional studies have demonstrated that CDH1 plays a critical role in lip and palate development during embryogenesis (Ghoumid 2017; Figueiredo 2019).

In the hereditary cancer genetics community, CDH1 is more commonly associated with hereditary diffuse gastric and lobular breast cancer syndrome (DGLBC). CDH1 variants linked to DGLBC are typically truncating mutations, resulting in a null allele. In contrast, CDH1 variants observed in individuals with BCDS are often missense mutations located in the EC1-EC2 linker region (amino acids 254-257) or exon 9 donor splice site variants (e.g., c.1320G>T, c.1320+1G>A, c.1320+1G>T, c.1320+1G>C, c.1320+5G>A) (Ghoumid 2017; Kievit 2018).

Historically, it was believed that individuals with BCDS-associated CDH1 missense variants were not at increased risk for DGLBC-associated cancers. This assumption was based on the absence of reported cancer cases in published BCDS families and epidemiological data from the CDH1 ClinGen Variant Curation Expert Panel (VCEP), which suggested that missense variants may not confer elevated cancer risk (Ghoumid 2017; Kievit 2018; Lee 2018).

However, a 2020 case report by LeBlanc et al. described a family with a known BCDS-associated CDH1 missense variant (c.768T>A, p.N256K), in which a 37-year-old male developed diffuse gastric cancer. This report raised concerns about potential cancer risks in individuals with BCDS-associated CDH1 variants and prompted questions regarding the need for endoscopic screening and other surveillance measures.

Currently, data regarding cancer risk in individuals with CDH1 variants and the BCDS phenotype are limited. The condition is rare, and affected individuals are often identified through exome sequencing due to multiple congenital anomalies. The interpretation of familial cancer risk is further complicated by a high rate of de novo mutations and limited family history.

To address these gaps, this registry aims to establish a centralized, international cohort of individuals with CDH1-associated BCDS. The goal is to better characterize the genotype-phenotype correlations, define the clinical spectrum, and assess the potential cancer risks associated with these variants.

ELIGIBILITY:
Inclusion Criteria:

* A documented pathogenic, likely pathogenic or a variant of uncertain significance in the CDH1 gene
* Clinical features that are diagnostic for, or suggestive of, BCDS (cleft lip and/or palate, eyelid anomalies, dental abnormalities, webbed toes, imperforate anus, etc)

Exclusion Criteria:

• Non-English-speaking individuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participation is not limited by location. There are two ways eligible patients can be referred:
  * Provider referral: The registry can be discussed with the potential study participant, and if they're interested, verbal permission can be obtained for our study team to reach out. With their consent, the study participant's name and preferred contact information can be sent to bcdsregistry@osumc.edu.
  * Self-referral: Potential study participants can express interest in study participation by visiting the registry website (https://redcap.link/BCDSregistry).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive characterization of the clinical phenotype associated with CDH1-associated blepharocheilodontic syndrome (BCDS) | 5 years
  Reporting of currently known clinical characteristics of CDH1-associated Blepharocheilodontic Syndrome (BCDS), including but not limited to cleft lip and/or palate, eyelid anomalies, dental abnormalities, webbed toes, and imperforate anus. The study will also document additional clinical features that may not have been previously reported in the literature, with the goal of expanding the phenotypic understanding of this rare condition.

SECONDARY OUTCOMES:
Development of evidence-based cancer surveillance recommendations for individuals with CDH1-assocaited blepharocheilodontic syndrome. | 10 years
  Personal and family cancer history will be collected and reviewed annually to evaluate potential cancer risks associated with CDH1 variants in individuals with blepharocheilodontic syndrome (BCDS). For participants who are of appropriate age and undergoing endoscopic surveillance as part of their routine medical care, relevant endoscopic and pathology reports will be obtained and analyzed to assess the presence and prevalence of signet ring cells, a hallmark of diffuse gastric cancer. This comprehensive data collection will support efforts to develop evidence-based cancer surveillance recommendations tailored to individuals with CDH1-associated BCDS.

CONTACTS AND LOCATIONS:
Overall Officials: Maegan E Roberts, MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be broadly shared. However, external requests for data access may be considered for use in downstream research protocols. All such requests must include an IRB-approved protocol and a formal application for data use. The BCDS Registry Advisory Board, comprising the Principal Investigator and at least one co-investigator, will review applications based on scientific merit and relevance, with input from a statistician as needed.
  For approved requests, data will be shared via a secure "data push," typically involving export from REDCap to a coded-limited file format. The individual responsible for data transfer will be certified as an honest broker under the OSUWMC Honest Broker Protocol. All studies using registry data will be conducted under separate IRB oversight.
Supporting Information: Study Protocol
Time Frame: Beginning after study accrual has reached 20 with no end date
Access Criteria: All research studies, whether internal or external to The Ohio State University, using data from the CDH1-associated BCDS Registry must be conducted under separate IRB approvals. Interested collaborators should email bcdsregistry@osumc.edu to request an Application for Use of Data. The application must include documentation of an IRB-approved protocol describing the proposed use of the data.

REFERENCES:
- [Background] Lee K, Krempely K, Roberts ME, Anderson MJ, Carneiro F, Chao E, Dixon K, Figueiredo J, Ghosh R, Huntsman D, Kaurah P, Kesserwan C, Landrith T, Li S, Mensenkamp AR, Oliveira C, Pardo C, Pesaran T, Richardson M, Slavin TP, Spurdle AB, Trapp M, Witkowski L, Yi CS, Zhang L, Plon SE, Schrader KA, Karam R. Specifications of the ACMG/AMP variant curation guidelines for the analysis of germline CDH1 sequence variants. Hum Mutat. 2018 Nov;39(11):1553-1568. doi: 10.1002/humu.23650. PMID 30311375
- [Background] Kievit A, Tessadori F, Douben H, Jordens I, Maurice M, Hoogeboom J, Hennekam R, Nampoothiri S, Kayserili H, Castori M, Whiteford M, Motter C, Melver C, Cunningham M, Hing A, Kokitsu-Nakata NM, Vendramini-Pittoli S, Richieri-Costa A, Baas AF, Breugem CC, Duran K, Massink M, Derksen PWB, van IJcken WFJ, van Unen L, Santos-Simarro F, Lapunzina P, Gil-da Silva Lopes VL, Lustosa-Mendes E, Krall M, Slavotinek A, Martinez-Glez V, Bakkers J, van Gassen KLI, de Klein A, van den Boogaard MH, van Haaften G. Variants in members of the cadherin-catenin complex, CDH1 and CTNND1, cause blepharocheilodontic syndrome. Eur J Hum Genet. 2018 Feb;26(2):210-219. doi: 10.1038/s41431-017-0010-5. Epub 2018 Jan 18. PMID 29348693
- [Background] Ghoumid J, Stichelbout M, Jourdain AS, Frenois F, Lejeune-Dumoulin S, Alex-Cordier MP, Lebrun M, Guerreschi P, Duquennoy-Martinot V, Vinchon M, Ferri J, Jung M, Vicaire S, Vanlerberghe C, Escande F, Petit F, Manouvrier-Hanu S. Blepharocheilodontic syndrome is a CDH1 pathway-related disorder due to mutations in CDH1 and CTNND1. Genet Med. 2017 Sep;19(9):1013-1021. doi: 10.1038/gim.2017.11. Epub 2017 Mar 16. PMID 28301459
- [Background] Figueiredo J, Melo S, Carneiro P, Moreira AM, Fernandes MS, Ribeiro AS, Guilford P, Paredes J, Seruca R. Clinical spectrum and pleiotropic nature of CDH1 germline mutations. J Med Genet. 2019 Apr;56(4):199-208. doi: 10.1136/jmedgenet-2018-105807. Epub 2019 Jan 19. PMID 30661051
- See also: CDH1-associated blepharocheilodontic syndrome (BCDS) registry website — https://redcap.link/BCDSregistry